CLINICAL TRIAL: NCT04899037
Title: Pilot Study to Evaluate the Long-term Chronic Care of Patients Who Could or do Utilize an Osseointegrated Device (OID)
Status: Recruiting | Type: Observational
Sponsor: University of South Florida (Other)
Collaborators: Oticon Medical (Industry)
Responsible Party: Principal Investigator, Victoria Sanchez (Williams), Principal Investigator, University of South Florida
Other Study IDs: STUDY001352
Record Dates: First submitted 2021-05-19; First posted 2021-05-24 (Actual); Last update posted 2025-10-28 (Actual); Status verified 2025-10

CONDITIONS: Hearing Loss, Conductive; Hearing Loss, Mixed; Deafness, Unilateral
Keywords: osseointegrated device; cognition; hearing loss; neurocognitive; BAHA; Ponto; Osseointegrated Bone-Conducting Hearing Protheses; Osia; Osseointegrated Auditory Device; Auditory Wellness
MeSH Terms: conditions — Hearing Loss, Conductive; Hearing Loss, Mixed Conductive-Sensorineural; Hearing Loss, Unilateral; Hearing Loss

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Osseointegrated Device Uptake: The participants in this group will be in the 18-85 year age range who have a hearing loss configuration that would benefit from an OID and choose to uptake an OID.
  Interventions: Other: No intervention
- Osseointegrated Device Non Uptake: The participants in this group will be in the 18-85 year age range and who a hearing loss configuration that would benefit from an OID but choose to not uptake an OID.
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — This is an observational study of participants that either choose or not choose to utilize an OID. This is not an intervention prescribed study, however, participants may choose uptake of standard of care intervention and obtain and utilize an OID. An OID is an FDA-approved device commonly recommended to patients with conductive, mixed, or singled-sided hearing loss. There is no experimental intervention evaluated in this study.

SUMMARY:
The primary objective of the study is to evaluate OID hearing intervention on cognition among patients who could vs. do utilize an OID. We will also evaluate the long-term effects of OID use on secondary outcomes measures (hearing performance, quality-of-life, social interaction, communication, physical functioning, etc)

DETAILED DESCRIPTION:
Hearing impairment is highly prevalent and independently associated with cognitive decline. Little is known about the various types, degrees, and configurations of hearing loss and how it relates to uptake of a hearing intervention and possible long-term benefits of using the intervention. The purpose of this study is to investigate the comparative effectiveness within an observational study design to determine the long-term effects of hearing intervention, in the form of osseointegrated devices (OID), among patients with either conductive, mixed, or single-sided hearing loss. Participants will be followed for 3 years (36 months) to answer the following aims:

Aim 1: To compare the effect of OID intervention versus no audiological intervention on rates of decline in global cognitive function (primary outcome measure) in 18-85 year-old well-functioning and cognitively-normal older adults with hearing loss. We hypothesize that there will be a significant difference in cognitive function between patients that utilized OID hearing intervention compared to no audiological intervention.

Secondary Aims: To compare the effect of OID intervention on secondary outcomes of hearing, social, mental, physical, and cognitive functioning. We hypothesize that there are significant differences in secondary outcomes between patients that utilized OID hearing intervention compared to no audiological intervention.

ELIGIBILITY:
Inclusion Criteria:

* age 18-85 years
* community dwelling
* residency: participants must plan to reside in the local area for the study duration.
* fluent English-speaker
* Audiometric hearing impairment: participants must have hearing configuration that could benefit from OID hearing intervention.
* Mini-Mental State Exam (MMSE) score > 23 for individuals with high-school degree or less; Mini-Mental State Exam (MMSE) score >25 for individuals with some college or more; participants must be at risk for cognitive decline the range quantified well by neurocognitive testing, and so must be free from more substantial cognitive impairment at baseline.
* willingness to participant and adhere to the protocol: participants must be willing and able to consent to participate in the study and be willing to commit to adhere to the study protocol for the duration of the study (3 years)

Exclusion Criteria:

* self-reported disability in >2 or more Activities of Daily Living (ADL)
* medical contraindication to use of OID; because OIDs will be the primary device used in the hearing intervention, participants with medical contraindications to OID use are excluded

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: adults age 18-85 years with an audiometric configuration (conductive or mixed hearing loss, single sided deafness) would could benefit from an OID hearing intervention
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2021-01-29 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Change from baseline to month 36 on Ensuring Speech Understanding Test scores, evaluating a participants ability to hear the examiner during the Neurocognitive Test Battery | Baseline and Month 36
  In this test, five sentences are read aloud to the participant by a research staff member, and the participant is asked to repeat back the sentence. Participants are scored on the number of target words repeated back correctly (3 target words/sentence). This test contains 2 trials, Trial 1 and Trial 2, with Trial 2 only being completed if the score on Trial 1 is below the specified criteria. The total score for Trail 1 is 1 (one target word repeated correctly) to 15 (all target words repeated correctly). If a participant's score is 12 or less on Trial 1, Trial 2 will be administered using a slightly louder tone. Trial 2 contains 15 target words and the same scoring criteria as Trail 1. If the score on Trial 2 is 12 or less, the examiner will use a slightly louder tone while administering the neurocognitive test battery. This test guards against poor speech understanding from hearing loss directly confounding administration of neurocognitive tests with auditory stimuli.
Change from baseline to month 36 on Mini Mental State Exam scores, evaluating cognitive function ability | Baseline and Month 36
  This test is a standardized instrument for screening a limited number of cognitive functions. The MMSE is used to exclude those with significant cognitive impairment at baseline, and as an outcome for tracking cognitive decline, and dementia. The MMSE is administered by interview and should be attempted in all participants. Scores range from 0 (no cognitive function questions answered correctly) to 30 (all cognitive function questions answered correctly).
Change from baseline to month 36 on Delayed Word Recall Test scores, evaluating verbal memory | Baseline and Month 36
  The DWRT is a measure of verbal memory that requires the participant to recall a list of 10 common nouns following a short delay. The participant is presented with a stimulus card for each of the 10 words. The examiner reads each word aloud, and asks the participant to repeat the word and use it in a sentence. This procedure is repeated, providing two exposures to the words. Following an approximate 5-minute delay, during which the (non-verbal) digit symbol substitution test (DSST) is given, the participant is asked to recall as many words as possible. Scores range from 0 (no words recalled correctly) to 10 (all words recalled correctly).
Change from baseline to month 36 on Digit Symbol Substitution Test scores, evaluating psychomotor speed and sustained attention | Baseline and Month 36
  The DSST is a measure of psychomotor speed and sustained attention and also serves as a nonverbal distractor task, interposed between learning and recall for the Delayed Word Recall Test (DWRT). The participant is asked to translate numbers (1-9) to symbols using a key provided at the top of the test form. The participant is provided with a pencil (without an eraser). Instructions are provided in a deliberate and slow pace. One point is given for each correctly drawn symbol completed within the 90-second time limit. Scores range from 0 (no symbols correctly drawn) to 93 (all symbols correctly drawn).
Change from baseline to month 36 on Incidental Learning Test scores, evaluating non-verbal recent memory | Baseline and Month 36
  The Incidental Learning Test was adapted from the WAIS-R NI and provides a non-verbal measure of recent memory. Following the Digit Symbol Substitution Test (DSST), the participant is presented with the Incidental Learning Template. The participant is asked to write down as many of the DSST symbols as he/she can remember, in any order. Next, the participant is asked to write down the number that was paired with each of the symbols from the DSST. Two scores are yielded: 1) Free Recall: total number of symbols recalled, regardless of pairing and 2) Pairing: number of correct symbols correctly paired with corresponding numbers. Scores for each range from 0 (no symbols recalled, no symbols correctly paired to corresponding numbers) to 9 (all symbols recalled, all symbols correctly paired to corresponding numbers).
Change from baseline to month 36 on Trail Making Test Part A (TMT A) scores, evaluating attention, sequencing, mental flexibility, visual search, and motor function | Baseline and Month 36
  The TMT A is a timed task in which participants connect numbers in sequence as quickly as possible. TMT measures attention, sequencing, mental flexibility, and visual search and motor function. In the TMT A, the participant is asked to draw a line and connect a series of numbers (from 1-25) as quickly as possible. Prior to the test part, the participant is given a sample test to demonstrate the task. The score for TMT A is the number of seconds required to complete the task. Scores range from 1 (1 second to connect all numbers) to 240 (240 seconds to connect all numbers). A maximum of 240 seconds (4 minutes) and 5 errors is allowed. If a participant makes 5 errors, the test is stopped even if the participant has not reached the 240 second limit, and a score of 240 seconds is given.
Change from baseline to month 36 on Trail Making Test Part B (TMT B) scores, evaluating attention, sequencing, mental flexibility, visual search, and motor function | Baseline and Month 36
  The TMT Part B is a timed task in which participants connect letters and numbers in sequence as quickly as possible. The TMT measures attention, sequencing, mental flexibility, and visual search and motor function. In the TMT B, the participant is asked to draw a line and connect a series of numbers and letters, alternating between a given number and letter (e.g., 1 to A, A to 2, 2 to B, B to 3, etc.) as quickly as possible. Prior to the test part, the participant is given a sample test to demonstrate the task. The score for TMT B is the number of seconds required to complete the task. Scores range from 1 (1 second to connect all numbers and letters) to 240 (240 seconds to connect all numbers and letters). A maximum of 240 seconds (4 minutes) and 5 errors is allowed. If a participant makes 5 errors, the test is stopped even if the participant has not reached the 240 second limit, and a score of 240 seconds is given.
Change from baseline to month 36 on Logical Memory I and II scores, evaluating immediate and delayed verbal recall | Baseline to Month 36
  The Logical Memory I and II provides a measure of immediate and delayed verbal recall for the number of ideas presented in two stories, which are read to the participant. Both stories are read to the participant, and after each story is presented, the participant is asked to recall as much of the story as possible. The Logical Memory I score is calculated as the average number of ideas recalled from Story A and B. Each story contains 25 scoring units, the maximum score is 25 (25+25/2). An approximate 20-minute delay follows, during which the remaining (non-memory) tests are administered. Following the delay period, the participant is again asked to recall the stories. The Logical Memory II score is calculated as the average number of story elements recalled from Story A and B. Scores range from 0 (no story elements correctly recalled) to 25 (all story elements correctly recalled).
Change from baseline to month 36 on Digit Span Backwards scores, evaluating attention and working memory | Baseline to Month 36
  The Digit Span Backwards is part of the Wechsler Memory Scale-Revised and provides a measure of attention and working memory. The participant is read a series of numbers progressively increasing in length from two to eight digits. After the numbers are read, the participant is asked to repeat the numbers in the reverse order. Two trials at each digit length are performed (i.e., 2 trials with 2 digits, 2 trials with 3 digits, etc.). The test is discontinued after two consecutive errors of the same length item. Scores range from 0 (no trails correctly repeated in reverse order) to 12 (all trials correctly repeated in reverse order).
Change from baseline to month 36 on Boston Naming Test scores, evaluating visual naming ability | Baseline to Month 36
  The Boston Naming Test assess visual naming ability using black-and-white drawings of common objects. For this study, the 30-item version used by the National Alzheimer's Coordinating Centers Uniform Data Set will be used. The participant is presented with a series of line drawings of objects and asked to name each object. The items become progressive more difficult based on their frequency of occurrence in the English language. A total score is calculated as the number of spontaneously produced correct responses. Scores may range from 0 (no object named correctly) to 30 (all objects named correctly).
Change from baseline to month 36 on Word Fluency Test scores, evaluating verbal functioning | Baseline to Month 36
  The Word Fluency Test is a measure of verbal functioning. In this task, the participant is asked to produce as many words as possible that begin with the letters F, A, and S within a time limit of 60 seconds for each letter, avoiding proper nouns, variations, plurals, and repetitions. The score is the total number of admissible words produced across letters, ranging from 0 (no words produced) to X (number of words produced).
Change from baseline to month 36 on Animal Naming Test scores, evaluating category fluency | Baseline to Month 36
  Animal Naming is a measure of category fluency (semantic association). Category fluency, and specifically animal naming, is part of the Boston Diagnostic Aphasia Examination, the Stanford-Binet test, and the CERAD. The participant is asked to name as many different animals as possible within a 60 second time limit. The score is given as the sum of all admissible names, from 0 (no animals named) to X (number of animals named).

SECONDARY OUTCOMES:
Change from baseline to month 36 on Oticon SSD Questionnaire (OSSDQ) ratings, evaluating why a patient wants to use OID hearing intervention | Baseline to Month 36
  The OSSDQ was developed by Oticon Medical as a brief instrument to capture reasons why a patient with single sided deafness may want to use OID hearing intervention. The OSSDQ is a self-administered questionnaire.
Change from baseline to month 36 on Tinnitus Functional Index (TFI) ratings, evaluating the intrusiveness of tinnitus in a participant's everyday life | Baseline to Month 36
  The Tinnitus Functional Index has eight subscales that address the intrusiveness of tinnitus, the sense of control the patient has, cognitive interference, sleep disturbance, auditory issues, relaxation issues, quality of life, and emotional distress. The subject will report (either directly onto the questionnaire in person, via web, or over the phone) answers to each of the 25 questions using a scale of 0 (tinnitus did not interfere) to 10 (tinnitus completely interfered).
Change from baseline to month 36 on Center for Epidemiological Studies Depression and Hopelessness Scale (CES-D) ratings, which screens for clinical depression | Baseline to Month 36
  The CES-D Short Form is a screening tool for identifying clinical depression, and is a self-administered questionnaire. Participants are asked to rate each item on a 3-point scale, 0 (hardly ever or never) to 2 (much or most of the time), on the basis of "how often you have felt this way during the past week."
Change from baseline to month 36 on Baecke Physical Activity Questionnaire (BPAQ) ratings, evaluating the frequency and duration of self report activities | Baseline to Month 36
  This is a self-administered questionnaire given to each participant that measures the frequency and duration of self-reported activities. This questionnaire asks about habitual physical activities including sport-related activities during leisure time, non-sport related physical activity during leisure time, and television viewing. Ratings range from A (least amount of physical activity) to E (highest amount of physical activity), with each question containing a different explanation for scores A-E based on the question asked.
Change from baseline to month 36 on Hearing Handicap Inventory for the Elderly (HHIE) ratings, evaluating the emotional and social impacts of hearing loss | Baseline to Month 36
  This is a self-administered screening questionnaire given to each participant to gather data on the perception of the impact of hearing loss. This questionnaire assesses the social and emotional impacts the participant perceives due to their hearing loss. Ratings range from 0 (No, hearing loss does not affect me) to 20 (Yes, hearing loss does affect me).
Change from baseline to month 36 on SF36 Health Survey (SF-36) ratings, evaluating health related quality of life | Baseline to Month 36
  The SF-36 Health Survey is a self-administered questionnaire that assesses health-related quality of life. It is a generic measure, as opposed to one that targets a specific age, disease, or treatment group. The SF-36 is the most widely-used health survey throughout the world because it is both brief and comprehensive, readily available, psychometrically-sound, and of proven usefulness in measuring health status and monitoring health outcomes. Eight domains of health can be estimated from the SF-36 (physical function, role limitations due to physical problems, social functioning, bodily pain, general mental health perception, role limitations due to emotional problems, emotional well-being, general health perception). Each domain is evaluated on a range of 0 (worst) to 100 (best) with a global median of 50.
Change from baseline to month 36 on Social Network Index (SNI) ratings, evaluating participant's social network | Baseline to Month 36
  The Cohen SNI is a self-administered questionnaire given to each participant to gather social network data. The Social Network Index evaluates two outcome variables: (1) Social Network Diversity - Number of social roles in which the participant had regular contact with for at least once every 2 weeks, and (2) People in Social Network -Total number of people with whom the participant had regular contact (at least once every 2 weeks). Examples of items include, "How many other relatives (other than your spouse, parents & children) do you feel close to?", "Do you attend any classes (school, university, technical training, or adult education) on a regular basis?", "Are you currently involved in regular volunteer work?", among others.
Change from baseline to month 36 in UCLA Loneliness Scale (UCLA - LS) ratings, evaluating participant's perception of loneliness | Baseline to Month 36
  This is a self-administered questionnaire given to each participant to gather loneliness data. This questionnaire measures subjective ratings of social isolation and loneliness (e.g. lacking companionship, feeling left out, and isolated from others, among others). Ratings range from 0 (never feeling what the question is asking) to 4 (always feeling what the question is asking).
Change from baseline to month 36 on Falls and Mobility ratings, measuring self reported physical ability, fatigue, and falls | Baseline to Month 36
  This is a self-administered questionnaire given to each participant to record living circumstances, self-reported physical ability, fatigue, and falls. Subjective ratings depend on the section being evaluated (e.g. no difficulty, never, 1 fall, do not remember).
Change from baseline to month 36 on Number of Hospitalizations | Baseline to Month 36
  This is a self-administered questionnaire given to each participant to record recent hospitalizations since the last time of study contact. Responses include Yes (hospitalized since last contact), or No (not hospitalized since last contact).

OTHER OUTCOMES:
Change from baseline to month 36 on the Audiometric Assessment, evaluating pure tone and speech audiometric abilities | Baseline to Month 36
  The audiometric diagnostic battery will be conducted by a trained audiology staff member for all participants. This assessment is standard of care. The battery includes otoscopy, tympanometry, pure tone audiometry, and speech audiometry (including word recognition testing in noise). The goal of this battery it to provide a diagnosis of hearing loss at the screening appointment, and then to monitor the participants hearing status during the study's time period.

CONTACTS AND LOCATIONS:
Overall Officials: Victoria Sanchez, Au.D, Ph.D, Principal Investigator — University of South Florida; Marsadi L Parliament, Au.D, Study Director — University of South Florida
Locations (1):
- Department of USF Health Otolaryngology; Auditory Rehabilitation & Clinical Trials Lab, Tampa, Florida, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Pickles JO. An introduction to the physiology of hearing. Bingley, UK: Emerald Group Publishing; 2008
- [Background] WHO. World Health Organization Prevention of Blindness and Deafness (PBD) Program. Prevention of Deafness and Hearing Impaired Grades of Hearing Impairment. <http://www.who.int/pbd/deafness/hearing_impairment_grades/en/index.html>.In.
- [Background] Lin FR, Niparko JK, Ferrucci L. Hearing loss prevalence in the United States. Arch Intern Med. 2011 Nov 14;171(20):1851-2. doi: 10.1001/archinternmed.2011.506. No abstract available. PMID 22083573
- [Background] Lin FR, Thorpe R, Gordon-Salant S, Ferrucci L. Hearing loss prevalence and risk factors among older adults in the United States. J Gerontol A Biol Sci Med Sci. 2011 May;66(5):582-90. doi: 10.1093/gerona/glr002. Epub 2011 Feb 27. PMID 21357188
- [Background] Chien W, Lin FR. Prevalence of hearing aid use among older adults in the United States. Arch Intern Med. 2012 Feb 13;172(3):292-3. doi: 10.1001/archinternmed.2011.1408. No abstract available. PMID 22332170
- [Background] Loughrey DG, Kelly ME, Kelley GA, Brennan S, Lawlor BA. Association of Age-Related Hearing Loss With Cognitive Function, Cognitive Impairment, and Dementia: A Systematic Review and Meta-analysis. JAMA Otolaryngol Head Neck Surg. 2018 Feb 1;144(2):115-126. doi: 10.1001/jamaoto.2017.2513. PMID 29222544
- [Background] Livingston G, Sommerlad A, Orgeta V, Costafreda SG, Huntley J, Ames D, Ballard C, Banerjee S, Burns A, Cohen-Mansfield J, Cooper C, Fox N, Gitlin LN, Howard R, Kales HC, Larson EB, Ritchie K, Rockwood K, Sampson EL, Samus Q, Schneider LS, Selbaek G, Teri L, Mukadam N. Dementia prevention, intervention, and care. Lancet. 2017 Dec 16;390(10113):2673-2734. doi: 10.1016/S0140-6736(17)31363-6. Epub 2017 Jul 20. No abstract available. PMID 28735855
- [Background] Rutherford BR, Brewster K, Golub JS, Kim AH, Roose SP. Sensation and Psychiatry: Linking Age-Related Hearing Loss to Late-Life Depression and Cognitive Decline. Am J Psychiatry. 2018 Mar 1;175(3):215-224. doi: 10.1176/appi.ajp.2017.17040423. Epub 2017 Dec 5. PMID 29202654
- [Background] Lin FR, Albert M. Hearing loss and dementia - who is listening? Aging Ment Health. 2014;18(6):671-3. doi: 10.1080/13607863.2014.915924. No abstract available. PMID 24875093
- [Background] Reed NS, Altan A, Deal JA, Yeh C, Kravetz AD, Wallhagen M, Lin FR. Trends in Health Care Costs and Utilization Associated With Untreated Hearing Loss Over 10 Years. JAMA Otolaryngol Head Neck Surg. 2019 Jan 1;145(1):27-34. doi: 10.1001/jamaoto.2018.2875. PMID 30419131
- [Background] Deal JA, Goman AM, Albert MS, Arnold ML, Burgard S, Chisolm T, Couper D, Glynn NW, Gmelin T, Hayden KM, Mosley T, Pankow JS, Reed N, Sanchez VA, Richey Sharrett A, Thomas SD, Coresh J, Lin FR. Hearing treatment for reducing cognitive decline: Design and methods of the Aging and Cognitive Health Evaluation in Elders randomized controlled trial. Alzheimers Dement (N Y). 2018 Oct 5;4:499-507. doi: 10.1016/j.trci.2018.08.007. eCollection 2018. PMID 30364572
- [Background] Tjellstrom A, Granstrom G. Long-term follow-up with the bone-anchored hearing aid: a review of the first 100 patients between 1977 and 1985. Ear Nose Throat J. 1994 Feb;73(2):112-4. PMID 8168443